CLINICAL TRIAL: NCT03320395
Title: Treatment of Ex-vivo Small Bowel Mucosa With a Dedicated Radiofrequency Ablation (SB-RFA) Catheter.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left the institution.
Sponsor: The Cleveland Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLA 16-032
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Angiodysplasia
MeSH Terms: conditions — Angiodysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Small bowel RFA treatment (Experimental): Five small bowel samples each of the duodenum, jejunum and ileum will be recruited treated.
  Interventions: Device: Small bowel RFA treatment

INTERVENTIONS:
Device: Small bowel RFA treatment — The samples will be spread and fixed using needles. The prototype RFA-SB ablation catheter will be applied by the PI as follows to each section of duodenum, jejunum and ileum.
  The treating paddle of the prototype RFA-SB catheter will be pushed on the small bowel mucosa exerting the same pressure that would be applied endoscopically.
  12 J/cm2 will be applied every time with a 20 second interval between applications to simulate clinical practice.
  There will be two single applications to two separate specimen sites. There will be two double applications to two separate specimen sites. There will be two triple applications to two separate specimen sites. There will be two quadruple applications to two separate specimen sites.

SUMMARY:
Gastrointestinal angiodysplasia (GIAD, a.k.a. angioectasia, arteriovenous malformations or AVM, and vascular ectasia) are mucosal or submucosal dilated blood vessels, usually multifocal, and a frequent cause of obscure GI bleeding, especially mid-small bowel hemorrhage.

Endoscopic treatment using argon plasma coagulation (APC) is popular but presents limitations as application of the therapy is not uniform, and passing the catheter repetitively through the enteroscope may not be possible. Despite endoscopic treatment rebleeding rates are high, between 25 to 50%.

An improvement in our ability to treat GIAD endoscopically is desirable. An ablation catheter would need to be easy to use repetitively through the enteroscope, be more maneuverable to direct treatment to the lesions, and also cover more area of intestinal mucosa per treatment compared to APC, and it should be low risk for damage to the healthy intestinal mucosa.

Radiofrequency ablation (RFA) may hold the answer. It's efficacy for treatment of superficial Barrett esophagus is undisputed, and it has recently been used with success to treat gastric antral vascular ectasia (GAVE) a condition which is remarkably similar to GIAD.

DETAILED DESCRIPTION:
Gastrointestinal angiodysplasia (GIAD, a.k.a. angioectasia, arteriovenous malformations or AVM, and vascular ectasia) are mucosal or submucosal dilated blood vessels lined by epithelium with no overlying mucosal lesion formed due to a combination of sub-mucosal vein obstruction, hypoxemia and neovascularization. It is a frequent cause of obscure GI bleeding, and the most common finding when evaluating mid-small bowel hemorrhage. It is also more common in patients with underlying valvular heart disease (especially aortic stenosis), end-stage renal disease, and von Willebrand disease (acquired or congenital). These lesions are usually multifocal as forty to 60% of the patients will have more than one About half stop bleeding spontaneously but at least a quarter of patients will suffer recurrent GI bleeding manifested by overt bleeding (melena or hematochezia), persistent fecal occult blood or persistent iron deficiency anemia.

Management includes endoscopic therapy, surgery, therapeutic angiography, and pharmacological treatment. Endoscopic therapy including thermal methods (multi-polar electrocoagulation, argon plasma coagulation, laser), injections (sclerosants, saline, epinephrine), and mechanical methods (hemostatic clips, band ligators) are widely used to treat all causes of GI bleeding including GIAD. Argon plasma coagulation (APC) is the preferred mode of endoscopic therapy for GIAD due to availability, relative ease of use, and a perceived superficial rather than deep depth of burn; however, studies have shown that depth of tissue injury can be substantial. APC therapy may not be uniform as adequacy and depth of ablation depends on the presence of debris, mucous or blood between the APC probe and tissue, and the ability to target the tissue in the presence of breathing, intestinal peristalsis, and scope position. The APC catheter can also bend during repeated insertions, a necessary maneuver to remove the burned tissue debris on the tip of the catheter which otherwise affects the argon plasma beam and this may terminally damage it.

Angioectasia rebleeding rates are high, at least 25 to over 50%. An improvement in our ability to treat small bowel GIAD is desirable. An ablation catheter would need to be easy to use repetitively through the enteroscope, be more maneuverable to direct treatment to the lesions, and also cover more area of intestinal mucosa per treatment compared to APC, and it should be low risk for damage to the healthy intestinal mucosa while treating GIAD.

Radiofrequency ablation (RFA) may hold the answer. It's efficacy for treatment of superficial Barrett esophagus is undisputed, and it has recently been used with success to treat gastric antral vascular ectasia (GAVE) a condition which is remarkably similar to GIAD.

This study will determine the depth of burn achieved on fresh and healthy small bowel explants using a dedicated small bowel RFA catheter at usual RFA settings.

ELIGIBILITY:
Inclusion Criteria:

* Understand and provide informed consent.
* All patients must be over 18 years of age, otherwise no age restrictions.
* Healthy small bowel tissue has cleared by pathology as tissue that would otherwise be discarded.
* Patients who are undergoing planned resection of the small bowel will be recruited until the study endpoints are met.

Exclusion Criteria:

* Inability to provide informed consent.
* Inability to isolate disease free section of small bowel or sufficient small bowel to perform SB-RFA treatment..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Depth of small bowel mucosa treatment | 3 months
  Study of the effect of RFA treatment on ex-vivo healthy small bowel mucosa including duodenum, jejunum, and ileum.

IPD SHARING:
Plan to Share IPD: No